CLINICAL TRIAL: NCT01708460
Title: Feasibility Study: Evaluation of the Ulthera® System for Lifting and Tightening the Buttocks and Thighs
Brief Title: Feasibility Study: Ulthera Treatment of the Buttocks and Thighs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULT-118
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2013-09

CONDITIONS: Skin Laxity
Keywords: Ulthera® System; Ultherapy™ Treatment; Ulthera, Inc.; Ultrasound treatment for skin tightening
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ulthera-treated subjects (Experimental): All enrolled subjects will receive one Ultherapy treatment to one side of the body in the lateral buttock region. Following study completion, subjects may elect to receive a balancing treatment to the other side of the body.
  Interventions: Device: Ulthera System Treatment

INTERVENTIONS:
Device: Ulthera System Treatment — Focused ultrasound energy delivered below the surface of the skin.
  Other Names: Ultherapy™

SUMMARY:
Up to 30 subjects will be enrolled. Enrolled subjects will receive an Ulthera® treatment to one side of the body, treating the lateral buttock region. Follow-up visits will occur at 90 and 180 days post-treatment. Study images will be obtained pre-treatment, immediately post-treatment, and at each follow-up visit.

DETAILED DESCRIPTION:
This is a prospective, single-center, pilot clinical trial to evaluate the efficacy of the Ulthera® System to improve buttock and thigh skin laxity. Global Aesthetic Improvement Scale scores and patient satisfaction questionnaires will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 30 to 65 years.
* Subject in good health.
* Skin laxity in the buttocks and thighs.
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated and/or weight loss through the follow-up period.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
* Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at Visit 1 and be willing and able to use an acceptable method of birth control (e.g., barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following conditions is documented on the medical history: a) Postmenopausal for at least 12 months prior to study; b) Without a uterus and/or both ovaries; or c) A bilateral tubal ligation at least six months prior to study enrollment.

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* BMI equal to or greater than 40.
* Excessive subcutaneous fat in the buttocks and thighs.
* Excessive skin laxity in the buttocks and thighs.
* Significant weight fluctuation (±10 lbs) in the past 6 months.
* Taking weight-loss medications/supplements.
* Surgical or non-surgical treatments to the target areas in the last 12 months, e.g., liposuction.
* Inability to understand the protocol or to give informed consent.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-12; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Overall lifting and tightening of the buttocks and thighs. | 90 days post-treatment
  As determined by a masked, qualitative assessment of photographs at three months post-treatment compared to baseline.

SECONDARY OUTCOMES:
Overall aesthetic improvement. | 90 and 180 days post-treatment.
  As determined by GAIS completed by the Investigator and subject.
Overall subject satisfaction. | 90 and 180 days post-treatment
  As determined by subjects' completion of a Patient Satisfaction Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: David Goldberg, MD, Principal Investigator — Skin Laser and Surgery Specialist of New York and New Jersey
Locations (1):
- Skin Laser and Surgery Specialist of New York and New Jersey, New York, New York, United States